CLINICAL TRIAL: NCT05081297
Title: Qigong Effects on Mental Health of People Under Relative Isolation
Brief Title: Qigong and Social Isolation: Mental Health Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Jorge Pereira Machado, Principal Investigator, Universidade do Porto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QgIsolationMentalHealth
Record Dates: First submitted 2021-09-23; First posted 2021-10-18 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Mental Health Wellness 1
Keywords: Qigong; Mental health; social isolation; Traditional vegetative biofeedback therapy
MeSH Terms: conditions — Psychological Well-Being; Social Isolation | interventions — Qigong

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qigong practitioner group (Experimental): This arm is the experimental group where qigong intervention is going to be applied to practitioners with experience
  Interventions: Other: Qigong
- No practice (No Intervention): This group has no intervention and acts as control
- Beginner Qigong practitioner group (Experimental): This arm is the experimental group where qigong intervention is going to be applied to practitioners with no experience.
  Interventions: Other: Qigong

INTERVENTIONS:
Other: Qigong — Qigong as a traditional chinese medicine technique, composed of several types of exercises: Baduanjin, taijiquan, yijinjing, baojiangong.
  Other Names: Traditional vegetative biofeedback therapy; Chikung; Taichi
  Arms: Beginner Qigong practitioner group; Qigong practitioner group

SUMMARY:
The objective of the study is to understand if Qigong may be useful in controlling the psychological state of participants in relative social isolation (during Covid-19 governmental imposed isolation procedures) The sessions are conducted live by the internet by a professional instructor-therapist with the duration of 2 months and a regular minimum of 2 sessions a week.

DETAILED DESCRIPTION:
The study's objective is to understand if Qigong may be helpful on the psychological state control of the participants in a relative state of isolation imposed by the government on the fight against Covid-19.

Data is gathered via the Mental Health Inventory (MHI) adapted to the Portuguese population to assess quantitative mental health scores and a simple structured interview to assess qualitative mental health benefits of Chikung (Qigong).

Qigong was the chosen technique to be studied as an intervention. Qigong is a Traditional Chinese Medicine therapeutic tool that has been studied for its several health benefits. As a traditional vegetative biofeedback therapy, Qigong can be useful for the maintenance of mental health of people with several conditions such as anxiety and depression, autism spectrum disorder and even conditions related to behavioral control.

* Group 1 was composed of Qigong practitioners (for at least 3 months).
* Group 2 was composed of participants who would receive the Qigong intervention (never practiced Qigong).
* Group 3 was composed of control participants (who would not receive the intervention).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Physical or mental disabilities or conditions that may aggravate when performing semi-supervised physical activity

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Psychological Well-being (Mental health Inventory (MHI) dimension) | T0 - Baseline week 0
  A higher score means a higher Psychological Well-being (0-100 score)
Psychological Well-being (Mental health Inventory (MHI) dimension) | T1 - 8 weeks
  A higher score means a higher Psychological Well-being (0-100 score)
Psychological Distress (Mental health Inventory (MHI) dimension) | T0 - Baseline week 0
  A higher score means a higher Psychological Distress (0-100 score)
Psychological Distress (Mental health Inventory (MHI) dimension) | T1 - 8 weeks
  A higher score means a higher Psychological Distress (0-100 score)

SECONDARY OUTCOMES:
Positive Affect (Mental health Inventory (MHI) dimension) | T0 - Baseline week 0
  A higher score means a higher Positive Affect (0-100 score)
Positive Affect (Mental health Inventory (MHI) dimension) | T1 - 8 weeks
  A higher score means a higher Positive Affect (0-100 score)
Emotional Ties (Mental health Inventory (MHI) dimension) | T0 - Baseline week 0
  A higher score means higher Emotional Ties (0-100 score)
Emotional Ties (Mental health Inventory (MHI) dimension) | T1 - 8 weeks
  A higher score means higher Emotional Ties (0-100 score)
Loss of emotional or behavioral control (Mental health Inventory (MHI) dimension) | T0 - Baseline week 0
  A higher score means a higher Loss of emotional or behavioral control (0-100 score)
Loss of emotional or behavioral control (Mental health Inventory (MHI) dimension) | T1 - 8 weeks
  A higher score means a higher Loss of emotional or behavioral control (0-100 score)
Anxiety (Mental health Inventory (MHI) dimension) | T0 - Baseline week 0
  A higher score means higher Anxiety levels (0-100 score)
Anxiety (Mental health Inventory (MHI) dimension) | T1 - 8 weeks
  A higher score means higher Anxiety levels (0-100 score)
Depression (Mental health Inventory (MHI) dimension) | T0 - Baseline week 0
  A higher score means higher Depression levels (0-100 score)
Depression (Mental health Inventory (MHI) dimension) | T1 - 8 weeks
  A higher score means higher Depression levels (0-100 score)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Machado, PhD, Study Director — ICBAS - Instituto de Ciências Biomédicas Abel Salazar; Lara Lopes, MSc, Principal Investigator — ICBAS - Instituto de Ciências Biomédicas Abel Salazar; Jorge M Rodrigues, BSc, Principal Investigator — ICBAS - Instituto de Ciências Biomédicas Abel Salazar
Locations (1):
- Instituto Português de Taichi e Chikung, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT05081297/Prot_SAP_ICF_000.pdf